CLINICAL TRIAL: NCT03798457
Title: Incidence and Prognostic Implication of Acute Cardiovascular Events in Patients Hospitalized for Community-acquired Pneumonia in Internal Medicine Units.The FADOI-ICECAP Study.
Brief Title: Incidence and Prognostic Implication of Acute CV Events in Patients Hospitalized for CAP in Internal Medicine Units.
Acronym: ICECAP
Status: Completed | Type: Observational
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: FADOI.06.2015
Record Dates: First submitted 2018-12-28; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Events
Keywords: Community-acquired pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CAP hospitalized in IM: Data of Patients with Community-acquired pneumonia (CAP) hospitalized in Internal Medicine Units will be collected for this study; no intervention is planned for this study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — In this study there is no intervention

SUMMARY:
FADOI-ICECAP is a observational, prospective, multicenter study involving 20-25 nationwide Units of Internal Medicine. The study foresees the participation of 26 Internal Medicine Operative Units, and for each of them a prospective registration of data relative to at least 50 patients admitted with CAP (in total, at least 1300 evaluable subjects) is foreseen.

DETAILED DESCRIPTION:
Phase 1 - Patients enrollment (October 2016 - February 2018) Each Investigator have recorded data concerning 50 patients. It will be collected general characteristics of patients, clinical parameters and conditions, diagnostic imaging and blood tests,

Phase 2 - Database review and validation (April 2018 - October 2018) The data collected will be analysed to process the endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Diagnosis of pneumonia defined by the presence on chest X-ray or CT-scan of lung of new infiltration associated with at least two of the following clinical features:

   * fever > 37.8°C
   * typical symptoms (dyspnea, productive cough, pain)
   * typical clinical signs on chest examination (crepitation, bronchial breathing, pleural effusion)
   * leukocytosis

Exclusion Criteria:

* patients with Hospital-Acquired Pneumonia (HAP) (i.e. those patients with pneumonia acquired in hospital more than 48 hours after admission)
* patients with tuberculosis in active phase
* patients with cystic fibrosis
* patients who refuse to participate in the study and/or to give the written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Community-acquired pneumonia (CAP) hospitalized in Internal Medicine Units
Sampling Method: Non-Probability Sample
Enrollment: 1266 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Incidence of CV events | 17 months
  To assess the cumulative incidence of well defined acute CV complications during hospitalization for CAP (index event).

SECONDARY OUTCOMES:
Mortality | 18 months
  To evaluate the impact on 30-day mortality of acute CV events occurred during hospitalization
Impact of acute CV events | 18 months
  To assess the impact of acute CV events occurred during hospitalization on the risk of hospital readmission within 30 days
Impact of CV events | 18 months
  To assess the impact of CV events on the length of hospitalization
Risk factor | 18 months
  To evaluate risk factors for the occurrence of acute CV events
Incidence of CV events in patients without history of heart failure, acute coronary syndrome, cerebrovascular disease, or clinically relevant arrhythmia | 18 months
  To evaluate the incidence of CV complications in the group of patients without history of heart failure, acute coronary syndrome, cerebrovascular disease, or clinically relevant arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Gussoni, MD, Study Director — Fadoi Foundation

REFERENCES:
- [Derived] Pieralli F, Vannucchi V, Nozzoli C, Augello G, Dentali F, De Marzi G, Uomo G, Risaliti F, Morbidoni L, Mazzone A, Santini C, Tirotta D, Corradi F, Gerloni R, Gnerre P, Gussoni G, Valerio A, Campanini M, Manfellotto D, Fontanella A; FADOI-ICECAP Study Group. Acute cardiovascular events in patients with community acquired pneumonia: results from the observational prospective FADOI-ICECAP study. BMC Infect Dis. 2021 Jan 25;21(1):116. doi: 10.1186/s12879-021-05781-w. PMID 33494707